CLINICAL TRIAL: NCT01502800
Title: A Phase 1 Dose Escalation and Pharmacodynamic Study of ARQ 761 (Beta-Lapachone) in Adult Patients With Advanced Solid Tumors
Brief Title: Clinical Trial of ARQ 761 in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU 042011-005; NCI-2011-03317 (Registry Identifier: CTRP)
Record Dates: First submitted 2011-10-18; First posted 2012-01-02 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Solid Tumors
Keywords: Metastatic; Unresectable; Recurrent advanced
MeSH Terms: conditions — Neoplasm Metastasis | interventions — beta-lapachone; RE1-silencing transcription factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Part 1 (ARQ 761) (Experimental): ARQ 761 (beta lapachone) will be given once a week. The same dose of ARQ761 each week for 4 weeks (1 cycle = 28 days). The total infusion time will be one (1) hour.
  Beginning dose level will be 195 mg/m2 and will increase until the maximum tolerated dose is defined. Seven dose levels that may be administered:
  1-195 mg/m2 2-390 mg/m2 3-450 mg/m2 4-550 mg/m2 5-660 mg/m2 6-800 mg/m2 7-1000 mg/m2
  Interventions: Drug: ARQ 761
- Part 2 Arm A (Experimental): The same dose of ARQ761 will be given each week for 8 weeks. The total infusion time will be 2 or 3 hours.
  Beginning dose level will be 390 mg/m2.
  Interventions: Drug: ARQ 761 Weekly Administration
- Part 2 Arm B (Experimental): ARQ 761 (beta lapachone) will be given bi-weekly for 8 weeks. The total infusion time may be either 2 or 3 hours.
  The beginning dose level will be 390 mg/m2.
  Interventions: Drug: Bi-Weekly Administration of ARQ 761
- Part 2 Arm C (Experimental): ARQ 761 (beta lapachone) will be given 2 consecutive weeks followed by one week of rest for 6 weeks. The total infusion time will be 2 or 3 hours.
  The beginning dose level will be 390 mg/m2.
  Interventions: Drug: Two Consecutive Weeks Administration of ARQ 761 with one week of rest

INTERVENTIONS:
Drug: ARQ 761 — ARQ 761 will be administered intravenously at a starting dose of 195 mg/m2 IV once weekly. Depending on toxicities observed, up to seven treatment cohorts will be enrolled with dose escalation occurring by doubling (first escalation) and 40% increments thereafter. If dosing is tolerated at all levels and pharmacokinetic data suggest continued escalation is warranted, additional dose levels will
  Other Names: Beta-Lapachone
  Arms: Part 1 (ARQ 761)
Drug: ARQ 761 Weekly Administration — If you decide to participate in this study ARQ 761 (beta lapachone) will be given to you through your vein once a week via a Portacath or Hickman line (a device that will make it easier to access your central vein that will be placed under your skin in your upper chest)
  You will receive the same dose of ARQ761 each week for 8 weeks. The total infusion time will be determined by your physician, it may be either 2 or 3 hours.
  The beginning dose level will be 390 mg/m2.
  Arms: Part 2 Arm A
Drug: Bi-Weekly Administration of ARQ 761 — If you decide to participate in this study ARQ 761 (beta lapachone) will be given to you through your vein bi-weekly via a Portacath or Hickman line (a device that will make it easier to access your central vein that will be placed under your skin in your upper chest)
  You will receive the same dose of ARQ761 bi-weekly for 8 weeks. The total infusion time will be determined by your physician, it may be either 2 or 3 hours.
  The beginning dose level will be 390 mg/m2.
  Arms: Part 2 Arm B
Drug: Two Consecutive Weeks Administration of ARQ 761 with one week of rest — If you decide to participate in this study ARQ 761 (beta lapachone) will be given to you through your vein once a week via a Portacath or Hickman line (a device that will make it easier to access your central vein that will be placed under your skin in your upper chest)
  You will receive the same dose of ARQ761 for 2 consecutive weeks followed by one week of rest for 6 weeks. The total infusion time will be determined by your physician, it may be either 2 or 3 hours.
  The beginning dose level will be 390 mg/m2.
  Arms: Part 2 Arm C

SUMMARY:
Primary Objective:

To determine the safety, tolerability and recommended Phase 2 dose (RP2D) of ARQ 761 administered intravenously.

Secondary Objectives:

To determine the pharmacokinetic profile of ARQ 761 To assess the preliminary anti-tumor activity of aRQ 761

DETAILED DESCRIPTION:
This is an open label, dose escalation study of (-)-trans-3-(5,6-dihydro-4H-pyrrolo [3,2,1-ij] quinolin-1-yl)-4(1Hindol-3-yl) pyrrolidine-2,5-dione (ARQ) 761. Drug administration regimen was designed in two parts.

Part I is a single-arm, non-randomized dose-escalation study. Part II is a multi-arm, randomized dose-escalation study. It is designed to establish the clinical tolerability and MTD of ARQ 761 and a recommended Phase 2 dose (RP2D). This is the first-in-human study with ARQ 761.

Part I ARQ 761 will be administered intravenously at a starting dose of 195 mg/m2 IV once weekly. A cycle for any patient already enrolled will consist of weekly administration of ARQ 761 with cycles repeated every 4 weeks (28 days).

Part II Alternate dosing regimen of ARQ 761 will be evaluated at a starting dose of 390 mg/m2. ARQ 761 will be administered intravenously at the assigned duration (2 h or 3 h) weekly, biweekly or for two consecutive weeks followed by one week of rest. Patient will be randomized to Arm A, B or C after enrollment.

Depending on toxicities observed, up to seven treatment cohorts will be enrolled with dose escalation occurring by doubling (first escalation) and 40% increments thereafter. If dosing is tolerated at all levels and pharmacokinetic data suggest continued escalation is warranted, additional dose levels will be considered. Patients enrolled and assessed for dose limiting toxicities (DLTs) will be eligible for intra-patient dose escalation.

Pharmacokinetic assessments will be performed on the first and the forth infusion days following the different regimen to maintain continuity among all treatment groups. Safety and tolerability of ARQ 761 will be assessed for the duration of study treatment. Evaluation of potential anti-tumor activity of ARQ 761 will be performed at regular intervals while patients remain on study. Dose escalation of ARQ 761 will proceed until the maximum tolerated dose or recommended Phase 2 dose is reached.

Intra-patient escalation from lower dose levels to successfully administered dose levels will be allowed. In order for patients at lower dose levels to be eligible for dose escalation, they must tolerate therapy without experiencing any DLT. In addition, prior to escalation, a complete cohort of three patients must have completed two cycles of therapy at the higher dose level without experiencing any DLTs. Patients receiving doses of ARQ 761 may be escalated a maximum of two times to the next consecutive cohorts.

Subjects will be enrolled according to a 3+3 dose escalation scheme. Treatment will be staggered such that the first patient treated at each dose level will receive his or her initial infusion at least 1 week prior to subsequent patients in the same cohort. At least 3 patients within a dose cohort must complete the first cycle of therapy prior to enrolling subjects at the next dose level.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have a confirmed solid tumor that is metastatic, unresectable or recurrent and for which standard curative or palliative measures do not exist or are no longer effective.
2. Prior and concurrent therapy:

   Chemotherapy: At least four weeks since prior cytotoxic chemotherapy or 6 weeks since nitrosoureas or mitomycin.

   Molecular targeted agents including monoclonal antibodies and tyrosine kinase inhibitors: At least two weeks since last therapy.

   Endocrine therapy: Subject may be remain on LHRH antagonist therapy for prostate cancer if tumor progression has been confirmed.

   Radiotherapy: At least 3 weeks since most recent radiotherapy. Other investigational therapy: At least four weeks since any other investigational therapy.

   Concurrent therapy: No other concurrent anticancer or investigational therapy permitted except as noted above.
3. Measurable disease is not required, but will be evaluated in each subject when possible.
4. Age ≥18 years
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
6. Life expectancy ≥ three months.
7. Central venous access, such as a Portacath or Hickman Line.
8. Pretreatment clinical laboratory parameters within 14 days
9. Availability of 10 unstained slides or paraffin-embedded tissue block from archived tumor specimen.
10. Subjects must be recovered from any toxicity related to prior anti-neoplastic therapy (to grade <1). Patients with CTCAE grade 2 or less sensory neuropathy or any grade alopecia are eligible.

Exclusion Criteria:

1. Subjects who have had cytotoxic chemotherapy or treatment with monoclonal antibodies within 4 weeks, radiotherapy within 3 weeks, or other molecular targeted therapies.
2. Subjects may not be receiving any other investigational agents.
3. Subjects with known untreated brain metastases. Subjects with known, treated brain metastases must be stable with no symptoms for four weeks.
4. Subjects receiving enzyme-inducing antiseizure drugs ("EIASD").
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, significant pulmonary disease (shortness of breath at rest or mild exertion), uncontrolled infection or psychiatric illness/social situations that would limit compliance with study requirements.
6. Pregnant women and breastfeeding should be discontinued.
7. Absence of central venous access for administration of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2011-12-29 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Patients will receive an average of 4 cycles of ARQ 761 (corresponding with a treatment cycle of 16 weeks).
  To determine the recommended Phase 2 dose (RP2D) of ARQ 761 administered intravenously.

SECONDARY OUTCOMES:
Pharmacokinetic profile of ARQ761 | Samples will be drawn from each subject during first and fourth infusion of study drug
  Serial venous blood samples will be drawn from each subject during first and fourth infusion of study drug to determine the plasma levels of ARQ761.If the same dose is not administered for the first and fourth infusion of study drug, Pharmacokinetics (PK) samples will only be collected after the first dose. PK samples to be collected at pre-infusion, 15min,30min, 55min (5 mins before end of infusion), 75 min, 2,4,6,h post infusion, 24h, 48h, and 168h

CONTACTS AND LOCATIONS:
Overall Officials: David E Gerber, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center - Simmons Cancer Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gerber DE, Beg MS, Fattah F, Frankel AE, Fatunde O, Arriaga Y, Dowell JE, Bisen A, Leff RD, Meek CC, Putnam WC, Kallem RR, Subramaniyan I, Dong Y, Bolluyt J, Sarode V, Luo X, Xie Y, Schwartz B, Boothman DA. Phase 1 study of ARQ 761, a beta-lapachone analogue that promotes NQO1-mediated programmed cancer cell necrosis. Br J Cancer. 2018 Oct;119(8):928-936. doi: 10.1038/s41416-018-0278-4. Epub 2018 Oct 15. PMID 30318513